CLINICAL TRIAL: NCT00060697
Title: Family Intervention to Promote Health in Children
Brief Title: A Mother's Role in Delaying Onset of Sexual Activity in Her Children
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 5R01HD39541-2; 5R01HD039541 (NIH)
Record Dates: First submitted 2003-05-09; First posted 2003-05-12 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-05

CONDITIONS: Child Behavior; Adolescent Behavior
Keywords: Sexual risk taking; Mother-child communication; Problem behaviors
MeSH Terms: conditions — Child Behavior; Adolescent Behavior; Problem Behavior

INTERVENTIONS:
Behavioral: Adolescent sexual activity education for mothers

SUMMARY:
The goal of this study is to enhance the mother's role in promoting avoidance of sexual risks and problem behaviors in 6- to 12-year-old children. Consenting mothers will attend a 10-session program designed to enhance the quality of mother-child communication, identify sexual risks, and increase parental monitoring and self-efficacy.

DETAILED DESCRIPTION:
This study will identify personal, parental, peer, and community factors that predispose children ages 6 to 12 to early initiation of sexual behavior or that foster resilience to sexual risk taking. The study will then evaluate an intervention designed to enhance resilience factors and reduce risk factors among 6- to 12-year-old children. The study will focus on the mother's role in promoting resilience to sexual risk taking.

During the first phase of the study, 300 children and their mothers will be asked to complete a one-time interview that includes an assessment of risk and resilience factors. Information from the interviews will be used to modify an intervention currently being used in another study of parent-adolescent pairs. The modified intervention will then be tested to determine the efficacy of the intervention in reducing risk and enhancing resilience among children in this age group.

In the second phase of the study, 296 children and their mothers will be randomized to either the intervention or control group. All mothers will complete a baseline interview. Mothers in the intervention group will attend 10 group sessions that include short presentations, discussions, media presentations (videotapes), and interactive exercises, including self-assessments, role plays, and games. The group sessions include content and skill development related to parenting, communication, sexuality, peer pressure, and school involvement. Mothers in the control group receive written information on diet and physical activity. The written materials are presented in a self-help format to increase physical activity; a cookbook contains low fat recipes designed especially for African American men and women living in the Atlanta, GA, area.

All participants complete follow-up interviews at 6 and 12 months after the baseline interview. Primary outcomes for mothers include measures of resilience and communication related to sexual issues. For children, outcomes include measures related to possible sexual situations.

ELIGIBILITY:
Inclusion Criteria

* Member of a participating community-based organization
* Child 6 to 12 years of age and biological mother/legal guardian
* Ability to read and comprehend English
* Willing to participate

Ages: 6 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1300
Dates: Start 2000-12; Study Completion 2005-05

CONTACTS AND LOCATIONS:
Overall Officials: Colleen K DiIorio, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States